CLINICAL TRIAL: NCT01142232
Title: Phase I/II Study of Oral Lenalidomide and High Dose Melphalan Supported by Autologous Peripheral Blood Stem Cell Infusion for Patients With Multiple Myeloma
Brief Title: Lenalidomide and High Dose Melphalan Followed by Autologous Stem Cell Transplant in Multiple Myeloma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Attaya Suvannasankha (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor-Investigator, Attaya Suvannasankha, Assistant Professor of Clinical Medicine, Indiana University
Organization: Indiana University (Other)
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1005-06; IUCRO-0290
Record Dates: First submitted 2010-06-10; First posted 2010-06-11 (Estimated); Results first posted 2019-10-22 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
Keywords: autologous stem cell transplantation
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide

STUDY DESIGN:
Intervention Model Description: All patients will receive melphalan 100 milligrams (mg) per meters squared (m2) intravenously day -2 and day -1. Phase I patients will be enrolled sequentially into one of dose levels below and administered the corresponding lenalidomide dose. The recommended phase II dose based on dose limiting toxicities observed in the phase I portion will be used for lenalidomide dosing in the phase II portion of the trial Dose level -1 Lenalidomide 25 mg daily day -7 to day +2, Dose level 1 Lenalidomide 50 mg daily day -7 to day +2, Dose level 2 Lenalidomide 75 mg daily day -7 to day +2, Dose level 3 Lenalidomide 100 mg daily day -7 to day +2, Dose level 4 Lenalidomide 150 mg daily day -7 to day +2,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Melphalan with lenalidomide (Experimental): Melphalan will be given on Day -2 and Day -1. Lenalidomide will be given from Day -7 to Day +2.
  Interventions: Drug: Lenalidomide plus Melphalan during autologous stem cell transplantation; Drug: Lenalidomide maintenance

INTERVENTIONS:
Drug: Lenalidomide plus Melphalan during autologous stem cell transplantation — Patients will receive a fixed dose of melphalan, while the dose of lenalidomide is escalated according to the protocol defined cohorts. Lenalidomide is given on day -7 to day +2, while intravenous melphalan is given on day -2 and -1. Lenalidomide dosing will be in the morning at approximately the same time each day.
Drug: Lenalidomide maintenance — Lenalidomide maintenance therapy will begin on Day +100 to Day +110 provided the protocol-defined criteria are met. The initial starting dose of lenalidomide during maintenance is 10 mg daily on Days 1-28 of each 28-day cycle.

SUMMARY:
This is a research study for newly diagnosed multiple myeloma or multiple myeloma has returned (relapsed). Multiple myeloma is a type of cancer that begins in white blood cells called plasma cells. Plasma cells make proteins that help fight infections. Current therapy for multiple myeloma includes high dose chemotherapy and autologous (patient's own cells) stem cell transplantation.

There will be two parts (or phases) to this study:

The purpose of the first part is to find the highest dose of a drug called lenalidomide (Revlimid®) that can be given in combination with high dose melphalan without causing severe adverse events.

The purpose of the second part is to find out the effects of this treatment (good and bad) on multiple myeloma patients.

DETAILED DESCRIPTION:
Lenalidomide is a drug that interferes with the development of tiny blood vessels that help tumors grow. Lenalidomide in combination with dexamethasone is approved by the Food and Drug Administration (FDA) for the treatment of relapsed multiple myeloma. It is also approved for the treatment of specific types of myelodysplastic syndrome (MDS), another blood cancer. Other research studies using lenalidomide in combination with other drugs in subjects with newly diagnosed multiple myeloma also show good response rate.

High dose melphalan is approved by the FDA and is commonly used in multiple myeloma treatment prior to stem cell transplantation. This combination of lenalidomide, high-dose melphalan and stem cell transplantation has not been studied in newly diagnosed and relapsed multiple myeloma, so it is considered experimental. In research studies, "experimental" refers to a drug or procedure that has undergone basic laboratory testing and received approval from the US Food and Drug Administration (FDA) to be tested in human subjects. A drug or procedure may be approved by the FDA for use in one disease or condition, but be considered experimental in other diseases or conditions.

In this study, lenalidomide will be given together with melphalan (chemotherapy) with the hope that more disease will be killed before the stem cell transplant. Three months after the transplant, patients will take lenalidomide again with the hope that this will help prolong the time when the disease is in remission.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Patients with diagnosis of multiple myeloma at any stage of disease undergoing high dose chemotherapy and stem cell transplantation.
* Phase II: Patients with myeloma undergoing a first high dose chemotherapy and stem cell transplantation after achieving at least stable disease following induction therapy. Any induction regimen prior to transplantation is allowed. No more than 2 prior lines of therapy prior to transplantation are allowed.
* All previous therapy not associated with peripheral blood stem cell transplant, including radiation, hormonal therapy, and surgery, must have been discontinued 4 weeks prior to treatment in this study.
* ECOG performance status of </= 2 at study entry
* Laboratory test results within protocol-specified ranges
* All study participants must be registered into the mandatory RevAssist® program, and be willing and able to comply with the requirements of RevAssist®
* Females of childbearing potential must have negative pregnancy test within 24 hours of first prescription for lenalidomide and must commit to either continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control.
* Able to take aspirin daily as prophylactic anticoagulation
* Subject must have the minimum stem cell dose of 5.0 x 10^6 CD34+ cells/kg collected.

Exclusion Criteria:

* Pregnant or breast feeding females
* History of intolerance or resistance to lenalidomide
* Known hypersensitivity to thalidomide
* The development of erythema nodosum if characterized by a desquamating rash while taking thalidomide or similar drugs.
* Known seropositive for or active viral infection with human immunodeficiency vrus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV). Patients who are seropositive because of hepatitis b virus vaccine are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-08-27 (Actual); Primary Completion 2015-11-06 (Actual); Study Completion 2019-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Attaya Suvannasankha, MD, Principal Investigator — Indiana University School of Medicine
Locations (1):
- IU Simon Cancer Center, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This protocol was based on enrolling up to 16 patients phase I and up to 46 patients in phase II. The study enrolled 60 patients with 16 in phase I and 44 in phase II.
Groups:
- Phase I, Dose Level 1: All patients will receive Melphalan 100 mg/m2 intravenously day -2 and day -1 and Lenalidomide 50 mg given daily day -7 to day +2
- Phase I, Dose Level 2: All patients will receive Melphalan 100 mg/m2 intravenously day -2 and day -1 and Lenalidomide 75 mg given daily day -7 to day +2
- Phase I, Dose Level 3: All patients will receive Melphalan 100 mg/m2 intravenously day -2 and day -1 and Lenalidomide 100 mg given daily day -7 to day +2
- Phase I, Dose Level 4; Phase II: All patients will receive Melphalan 100 mg/m2 intravenously day -2 and day -1 and Lenalidomide 150 mg given daily day -7 to day +2
Period: Overall Study
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase II
Started | 3 | 4 | 3 | 6 | 44
Completed | 0 | 0 | 0 | 1 | 10
Not Completed | 3 | 4 | 3 | 5 | 34
Not completed — Adverse Event | 1 | 2 | 1 | 0 | 4
Not completed — Death | 0 | 0 | 0 | 0 | 1
Not completed — Disease Progression | 2 | 0 | 1 | 2 | 12
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 3
Not completed — Physician Decision | 0 | 1 | 0 | 2 | 10
Not completed — Alternative Therapy | 0 | 1 | 1 | 0 | 1
Not completed — Off Trt for other complicating disease | 0 | 0 | 0 | 0 | 1
Not completed — Noncompliance | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase II | Total
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 44 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 3 | 5 | 34 | 45
  >=65 years | 1 | 3 | 0 | 1 | 10 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (7.3) | 63.0 (11.7) | 56.1 (10.8) | 56.6 (9.1) | 58.6 (8.4) | 58.7 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1 | 1 | 13 | 16
  Male | 2 | 4 | 2 | 5 | 31 | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 3 | 6 | 43 | 59
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 1 | 4 | 5
  White | 3 | 4 | 3 | 5 | 38 | 53
  More than one race | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Number of Patients With Dose Limiting Toxicity
Description: The number of patients who had a DLT during the dose finding portion (Phase I) of the trial for the safety of lenalidomide when used in combination with high dose melphalan in the setting of autologous stem cell transplantation in patients with multiple myeloma.
Time Frame: up to 1 month
Population: All Phase I patients receiving at least one dose of study drug and having at least one evaluable post-baseline visit (16 patients)
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4
Number analyzed (Participants) | 3 | 4 | 3 | 6
Participants | 0 | 0 | 0 | 0

2. Primary Outcome: Phase II: Overall Response Rate
Description: Evaluate the overall response rate of patients receiving therapy. Patients are considered as having a response if their overall response is Partial Response or better (CR+sCR+VGPR+PR). The percentage of patients achieving this and the exact 95% confidence interval will be calculated. Responses will be defined using the response criteria determined by the International Working Group for Multiple Myeloma (CR= Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and 5% plasma cells in bone marrow; sCR=CR as defined above plus normal FLC ratio and absence of clonal cells in bone marrow by immunohistochemistry or immunoflurorescence; VGPR=Serum and urine M-component detectable by immunofixation but not on electrophoresis or 90% or greater reduction in serum M-component plus urine M-component<100 mg per 24 h; PR=>=50% reduction of serum M-protein and reduction in 24-h urinary M-protein by >=90% or to <200mg per 24 h).
Time Frame: up to 5 years
Population: All Phase II patients who received at least one dose of study drug and had at least one evaluable post-baseline visit
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 40
percentage of participants | 87.5 [73.2 to 95.8]

3. Secondary Outcome: Phase II: Treatment-Related Adverse Events Grade 3 or Higher
Description: Number of unique patients who had a treatment-related (possible, probable or definite) adverse events that were graded 3 or higher.
Time Frame: up to 5 years
Population: All Phase II patients who received treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase II
Number analyzed (Participants) | 44
Participants | 18

ADVERSE EVENTS:
Time Frame: up to 5 years
Arm/Group | Phase I, Dose Level 1 | Phase I, Dose Level 2 | Phase I, Dose Level 3 | Phase I, Dose Level 4 | Phase II
Serious Adverse Events (participants affected / at risk) | 0/3 | 1/4 | 2/3 | 3/6 | 11/44
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6 | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose Level 1 (N=3) | Phase I, Dose Level 2 (N=4) | Phase I, Dose Level 3 (N=3) | Phase I, Dose Level 4 (N=6) | Phase II (N=44)
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Colonic obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1 | 1 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0
Infections and infestations - Other (Infections and infestations) | 0 | 1 | 0 | 1 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1 | 1
Upper respiratory infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 1
Investigations - Other (Investigations) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 0 | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I, Dose Level 1 (N=3) | Phase I, Dose Level 2 (N=4) | Phase I, Dose Level 3 (N=3) | Phase I, Dose Level 4 (N=6) | Phase II (N=44)
Anemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 0 | 2 | 12
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 2
Cardiac disorders - Other (Cardiac disorders) | 0 | 0 | 0 | 1 | 2
Chest pain - cardiac (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
Ear and labyrinth disorders - Other (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 4
Hearing impaired (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 2
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 3
Eye disorders - Other (Eye disorders) | 0 | 1 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 1 | 0
Retinal detachment (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 12
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 1 | 3 | 25
Diarrhea (Gastrointestinal disorders) | 3 | 2 | 3 | 6 | 39
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 7
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 24
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 6 | 39
Oral dysesthesia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 1 | 4 | 18
Chills (General disorders) | 1 | 0 | 0 | 1 | 2
Edema limbs (General disorders) | 0 | 1 | 3 | 4 | 14
Fatigue (General disorders) | 3 | 3 | 3 | 6 | 32
Fever (General disorders) | 0 | 1 | 2 | 4 | 22
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 4
General disorders and administration site conditions - Other (General disorders) | 0 | 0 | 0 | 0 | 4
Injection site reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Localized edema (General disorders) | 0 | 0 | 0 | 1 | 2
Malaise (General disorders) | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 3
Pain (General disorders) | 0 | 3 | 1 | 3 | 20
Bronchial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 2
Infections and infestations - Other (Infections and infestations) | 0 | 3 | 1 | 3 | 8
Lung infection (Infections and infestations) | 0 | 1 | 0 | 1 | 7
Sinusitis (Infections and infestations) | 2 | 0 | 1 | 0 | 6
Skin infection (Infections and infestations) | 1 | 2 | 0 | 2 | 3
Upper respiratory infection (Infections and infestations) | 2 | 2 | 2 | 3 | 15
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 4
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 4 | 13
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1 | 3 | 6
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 4 | 15
Blood bilirubin increased (Investigations) | 1 | 2 | 2 | 4 | 16
Creatinine increased (Investigations) | 1 | 1 | 0 | 4 | 8
INR increased (Investigations) | 0 | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 2 | 3 | 0 | 2 | 10
Platelet count decreased (Investigations) | 1 | 2 | 0 | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2 | 12
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 3 | 2 | 0 | 0 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 2 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 1 | 3 | 16
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 2 | 3
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 4 | 11
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 1 | 1 | 2 | 8
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 1 | 4
Dysphasia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 2 | 8
Neuralgia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Paresthesia (Nervous system disorders) | 0 | 1 | 0 | 1 | 2
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 1 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 2 | 2 | 5 | 16
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 0 | 0 | 1 | 3
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 4
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 1 | 5
Insomnia (Psychiatric disorders) | 1 | 2 | 0 | 1 | 10
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 1
Urinary urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 2
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 1 | 4 | 13
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0 | 3 | 12
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 3
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 2 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 2
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 1
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 4
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 1 | 3 | 14
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 5
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 4
Hypotension (Vascular disorders) | 0 | 1 | 3 | 0 | 5
Superficial thrombophlebitis (Vascular disorders) | 0 | 0 | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 1 | 0 | 0 | 1
Vascular disorders - Other (Vascular disorders) | 1 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes